CLINICAL TRIAL: NCT04008329
Title: A Registered Cohort Study on Amyotrophic Lateral Sclerosis
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ning Wang, MD., PhD., Professor, First Affiliated Hospital of Fujian Medical University
Other Study IDs: MRCTA,ECFAH of FMU [2019]191
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; natural history; genetics; prognostic factors
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a kind of motor neuron degeneration disorder without effective therapy. This registered cohort study will provide further insights into the clinical course of ALS, and investigate disease-relative risk factors and the genetic background of Chinese ALS patients.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is the most common form of motor neuron disease (MND), which is characterized with highly clinical heterogeneity and no effective treatment is available now. The purpose of this registered cohort is to observe the natural history of ALS patients in China, and then identify some factors correlated with disease progression. Besides, ALS-related gene mutations will be screened and explore novel disease causing gene as well.

ELIGIBILITY:
Inclusion Criteria:

* Amyotrophic Lateral Sclerosis patients fulfilling the El Escorial criteria (including definite, probable and possible)
* Progressive muscular atrophy
* Primary lateral sclerosis
* Progressive bulbar palsy

Exclusion Criteria:

* History of serious head trauma or neuropsychiatric disease
* Decline to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ALS patients who are diagnosed in the First Affiliated Hospital of Fujian Medical University
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2059-07 (Estimated)

PRIMARY OUTCOMES:
Age at death | 10 years
  the time when patient die
Age of endotracheal intubation or tracheotomy | 10 years
  the time for the patient accepted endotracheal intubation or tracheotomy

CONTACTS AND LOCATIONS:
Overall Officials: Ning Wang, MD,PhD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Neurology, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Liu K, Guo Q, Ding Y, Luo L, Huang J, Zhang Q. Alterations in nasal microbiota of patients with amyotrophic lateral sclerosis. Chin Med J (Engl). 2024 Jan 20;137(2):162-171. doi: 10.1097/CM9.0000000000002701. Epub 2023 Jul 21. PMID 37482646